CLINICAL TRIAL: NCT04776512
Title: Lumbar Erector Spinae Plane Block Versus Classic Epidural Analgesia in Labor
Brief Title: Erector Spinae Plane Block Versus Classic Epidural Analgesia in Labor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor head of anesthesia and intensive care department, Mongi Slim Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESP versus Epidural analgesia
Record Dates: First submitted 2021-02-23; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Analgesia in Labor
Keywords: analgesia, vaginal delivery, ESP, EPIDURAL
MeSH Terms: conditions — Agnosia | interventions — Analgesia, Epidural

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural Analgesia (Experimental): Patients of this group Will receive an epidural analgesia through a lumbar epidural catheter
  Interventions: Procedure: Epidural Analgesia
- ESP Block (Experimental): Bilateral ESP block performed at the level of the 3 rd Lumbar transverse process.
  Interventions: Procedure: ESP Block With Bupivacain

INTERVENTIONS:
Procedure: ESP Block With Bupivacain — bilateral lumbar ESP block using 0.375% Bupivacain
  Arms: ESP Block
Procedure: Epidural Analgesia — Continuous Lumbar Epidural analgesia With 0,125% Bupivacain+0,25 mcg/ml Sufentanil
  Arms: Epidural Analgesia

SUMMARY:
Prosepective,Randomized, controlled study enrolling full termed parturients admitted for vaginal delivery.

At the sencond stage of labor: 3cm of cervix dilatation, patients will be randomized in 2 groups:

* ESP group: patients will receive ultrasound guided, bilateral ESP Block performed at the level of the 3 rd Lumbar transverse process.
* Epidural Analgesia Group: Patients will have a classic lumbar continuous epidural analgesia.

DETAILED DESCRIPTION:
Prosepective,Randomized, controlled study enrolling full termed parturients admitted for vaginal delivery.

At the sencond stage of labor: 3cm of cervix dilatation, patients will be randomized in 2 groups:

* ESP group: patients will receive ultrasound guided, bilateral ESP Block performed at the level of the 3 rd Lumbar transverse process.
* Epidural Analgesia Group: Patients will have a classic lumbar continuous epidural analgesia.

For the first group: 20 ml of 0,375% isobaric Bupivacain solution will be injected bilaterally under ultrasound direct vision.

Concerning the second group, patients will have a continuous injection of 0,125% Bupivacain solution associated to 0,25 mcg of Sufentanil/ml through an epidural catheter in the L3-L4 or L4-L5 intervertebral space.

For the 2 groups, analgesia will be assessed during all the labor period hourly using the Visual Analog pain Score (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Full termed parturients admitted for vaginal delivery
* singleton pregnancy
* No contraindications to perimedullar analgesia techniques

Exclusion Criteria:

* Indication to Cesarean section during labor period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — full termed parturients
Enrollment: 50 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Analgesia during labor | change in VAS score 1 hour after the beginning of labor
  analgesia assessed using VAScore

IPD SHARING:
Plan to Share IPD: No